CLINICAL TRIAL: NCT04294329
Title: Pre-emptive Quadratus Lumborum Block for Laparoscopic Bariatric Surgery.A Prospective Randomizes Controlled Study.
Brief Title: Pre-emptive Quadratus Lumborum Block for Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Walid Nofal, Clinical professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU R 18/2017
Record Dates: First submitted 2020-02-14; First posted 2020-03-04 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pain; Postoperative
Keywords: Quadratus lumborum block; laparoscopic bariatric surgery
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Quadratus lumborum block with bupivacaine (Experimental): After induction of anesthesia a QLB (quadratus lumborum block) will be performed by using ultrasound machine where a solution of 0.25% bupivacaine 0.2 ml /kg (lean body weight) is used on each side with care not to exceed the toxic dose.
  Interventions: Procedure: US-guided Quadratus lumborum block.; Drug: Bupivacaine
- Group Quadratus lumborum block with saline (Placebo Comparator): After induction of anesthesia a QLB (quadratus lumborum block) will be performed by using ultrasound machine.A volume of 0.2ml/kg normal saline will given for each side.
  Interventions: Procedure: US-guided Quadratus lumborum block.; Drug: Saline

INTERVENTIONS:
Procedure: US-guided Quadratus lumborum block. — Performance of quadratus lumborum block using ultrasound machine to relieve pain after bariatric surgery
Drug: Bupivacaine — Bupivacaine
  Arms: Group Quadratus lumborum block with bupivacaine
Drug: Saline — normal saline
  Arms: Group Quadratus lumborum block with saline

SUMMARY:
The purpose of this study was to determine the effectiveness of pre-emptive Quadratus lumborum block on intra, postoperative pain assessment and opioid requirements in laparoscopic bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

Patients included in this study are

* Both genders
* Age between 18-50 years
* Those undergoing laparoscopic bariatric surgery (as laparoscopic sleeve gastrectomy or gastric bypass).
* BMI ≥ 35 Kg/m2 with comorbidity or ≥ 40 Kg/m2 without comorbidity.

Exclusion Criteria:

Patients excluded from this study were

* those with obstructive sleep apnoea and/or Pickwickian syndrome.
* if the laparoscopy procedure was converted to laparotomy.
* patients suffering from known coagulation defects.
* known hypersensitivity to bupivacaine, or those with contraindication to the use of NSAIDS.
* Presence of sepsis at the site of injection.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain severity | 24 hours postoperatively
  Assessment of analgesia intraoperatively and for the first 24 hours postoperatively using the numerical ratingscale (NRS)score .The scale ranges from 0 to 10 where 0 indicates no pain and 10 indicates the worst pain imaginable.

SECONDARY OUTCOMES:
Intraoperative hemodynamics | 24 hours postoperatively
  Mean arterial pressure (MAP) in mmHg.
Postoperative analgesic needs | 24 hours postoperatively.
  Time to first analgesic requirement in hours
Total dose of opioids | 24 hours postoperatively.
  Total dose of opioids received in mg

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S. Omran, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Ain Shams University; Doaa M. Kamal El-Din, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Ain Shams Unive; Walid H. Nofal, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Ain Shams Unive
Locations (1):
- Anesthesiology department, Faculty of Medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No